CLINICAL TRIAL: NCT01583621
Title: Vitamin D Supplementation in Overweight/Obese African American Adults and Youth (D-SUNNY)
Acronym: D-SUNNY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Yanbin Dong, Professor, Department of Pediatrics, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: pro#00000051
Record Dates: First submitted 2012-04-03; First posted 2012-04-24 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (4):
- Placebo (No Intervention): Placebo group
- Supplementation arm 1 (Experimental): cholecalciferol 18000 U/month for 4 months
  Interventions: Dietary Supplement: Cholecalciferol
- supplementation arm 2 (Experimental): cholecalciferol 60000 U/month for 4 months
  Interventions: Dietary Supplement: Cholecalciferol
- Supplementation arm 3 (Experimental): cholecalciferol 120000 U/month for 4 months
  Interventions: Dietary Supplement: Cholecalciferol

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — The participants will be randomized into one of the four groups. Group 0 will be placebo group, group 1 will receive monthly supervised dose of 18,000 IU (equivalent to 600 IU/day), group 2 will receive monthly supervised dose of 60,000 IU(equivalent to 2000 IU/day), and group 3 will receive 120,000 IU (equivalent to 4000 IU/day) vitamin D3 supplementation for 4 months (16 weeks).
  Arms: Supplementation arm 1; Supplementation arm 3; supplementation arm 2

SUMMARY:
Primary Specific Aim 1: To compare the dose-responsive effects of vitamin D3 supplementations on 25(OH) D, parathyroid hormone (PTH), and serum/urine calcium.

Primary Specific Aim 2: To compare the dose-responsive effects of vitamin D3 supplementations on non-invasive vascular measures including pulse wave velocity (PWV), flow-mediated dilation (FMD), carotid arterial compliance (CAC), carotid Intima-Media Thickness (cIMT), and 24-hours Ambulatory Blood Pressure (ABP) monitoring as well as casual BP.

ELIGIBILITY:
Inclusion Criteria:

1. African-Americans (blacks)
2. Age 13-45
3. Overweight/obese (BMI ≥ 85th percentile for their age and gender for age 13-17 and BMI ≥ 25 kg/m2 for age 18-45)
4. Relatively healthy (no medical history of any heart, lung, endocrine or malignant disorder)
5. Non pregnant
6. Not on any medication or vitamin supplements that can influence the study outcomes
7. Serum 25 hydroxy Vitamin D (25[OH] D) levels ≤ 20 ng/ml (50 nmol/L) at the time of screening

Exclusion Criteria:

1. Not meeting any one or more of the above criteria
2. Females who become pregnant/test positive on urine pregnancy test during the screening or any of the testing visits
3. Anyone who is taking any multivitamin supplements that contains vitamin D

Ages: 13 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 74 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Cardiovascular phenotypes | 16 weeks
  Will be using non-invasive vascular measures including pulse wave velocity (PWV), flow-mediated dilation (FMD), carotid arterial compliance (CAC), carotid Intima-Media Thickness (cIMT), and 24-hours Ambulatory Blood Pressure (ABP) monitoring.
Primary outcome 1 dose-responsive effects of vitamin D3 supplementations | 16 weeks
  To compare the dose-responsive effects of vitamin D3 supplementations on 25(OH) D, parathyroid hormone (PTH), and serum/urine calcium.
Primary Outcome 2 dose-responsive effects of vitamin D3 supplementations | 16 weeks
  To compare the dose-responsive effects of vitamin D3 supplementations on non-invasive vascular measures including pulse wave velocity (PWV), flow-mediated dilation (FMD), carotid arterial compliance (CAC), carotid Intima-Media Thickness (cIMT), and 24-hours Ambulatory Blood Pressure (ABP) monitoring as well as casual BP.

CONTACTS AND LOCATIONS:
Overall Officials: Yanbin Dong, MD, PhD, Principal Investigator — Augusta University
Locations (1):
- Georgia Prevention Institute, Augusta, Georgia, United States

REFERENCES:
- [Derived] Bhagatwala J, Zhu H, Parikh SJ, Guo DH, Kotak I, Huang Y, Havens R, Pham M, Afari E, Kim S, Cutler C, Pollock NK, Dong Y, Raed A, Dong Y. Dose and time responses of vitamin D biomarkers to monthly vitamin D3 supplementation in overweight/obese African Americans with suboptimal vitamin d status: a placebo controlled randomized clinical trial. BMC Obes. 2015 Jul 4;2:27. doi: 10.1186/s40608-015-0056-2. eCollection 2015. PMID 26217542